CLINICAL TRIAL: NCT01010945
Title: A Phase Ib Study of Erlotinib in Combination With Gemcitabine and Nab-Paclitaxel in Patients With Previously Untreated Advanced Pancreatic Cancer
Brief Title: Erlotinib, Gemcitabine and Nab-Paclitaxel in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-774-108; 09PAN01 (Other: Criterium Inc.)
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Advanced Pancreatic Cancer
Keywords: erlotinib; nab-paclitaxel; gemcitabine; Adenocarcinoma; Advanced Pancreatic Cancer; Phase 1b
MeSH Terms: conditions — Adenocarcinoma | interventions — Erlotinib Hydrochloride; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- erlotinib, gemcitabine, nab-paclitaxel (Experimental): Patients receive the following treatment in 28-day cycles: 1) erlotinib: orally once daily from days 1 through 28 continuous dosing; 2) gemcitabine (following nab-paclitaxel): intravenously over 30 minutes on days 1, 8 and 15 every 28 days; and 3) nab-paclitaxel: intravenously over 30 minutes on days 1, 8 and 15 every 28 days.
  Interventions: Drug: erlotinib; Drug: gemcitabine; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: erlotinib — administered orally
  Other Names: Tarceva; OSI-774
Drug: gemcitabine — administered intravenously
Drug: nab-paclitaxel — administered intravenously

SUMMARY:
This is a phase 1b study to evaluate the combination of gemcitabine and Tarceva (erlotinib) and nab-paclitaxel in patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
This is a single-arm, phase 1b study to determine the maximum tolerated dose (MTD) of the combination of erlotinib (daily), gemcitabine (weekly), nab-paclitaxel (weekly) in patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1
* Predicted life expectancy of >= 12 weeks
* Previous surgery
* Histologically or cytologically confirmed, measurable, locally advanced, unresectable or metastatic pancreatic adenocarcinoma
* No prior therapy for pancreatic cancer
* Adequate organ and marrow function

  * Absolute neutrophil count >= 1.5 x 10^9/L
  * Platelets >= 100 x 10^9/L
  * Total bilirubin <= institutional upper limits of normal
  * AST (SGOT)/ALT(SGPT) <= 2 x institutional upper limits of normal
  * Serum creatinine <= 1.5 x upper limits of normal
* Negative pregnancy test
* Informed consent
* Patient must agree not to smoke while on study

Exclusion Criteria:

* Significant history of cardiac disease unless the disease is well controlled
* Active or uncontrolled infections or serious illness or medical conditions that could interfere with the patient's ongoing participation in study
* History of any psychiatric condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent
* History of smoking within the previous 14 days before enrollment or positive cotinine test at baseline
* Pregnant or breast-feeding females
* Symptomatic brain metastases that are not stable, that require steroids, that are potentially life-threatening, or that have required radiation within the last 14 days
* History of allergic reactions attributed to compounds of similar chemical or biological composition to the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-02-03 (Actual); Primary Completion 2012-01-25 (Actual); Study Completion 2012-01-25 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Monthly (to a maximum of 12 months)

SECONDARY OUTCOMES:
Safety of drug combination assessed through dose limiting toxicities (DLTs) | 1 month
Safety of drug combination assessed through Adverse Events (AEs) | Monthly (to a maximum of 12 months)
Evaluate erlotinib Pharmacokinetic (PK) trough concentrations (C24h) | Days 29 (Cycle 2, Day 1) and 30
Objective Response Rate | Monthly (to a maximum of 12 months)
  Response will be based on the RECIST v1.1 criteria. Patients with partial and complete response will be classified as "responders".
Progression Free Survival (PFS) | Monthly (to a maximum of 12 months)
  PFS will be calculated as the time from start of treatment until disease progression or death; patients who are still alive and free of progression at their last follow-up will be censored at that time.
Overall Survival | Monthly (to a maximum of 12 months)
  Survival will be calculated as the time from start of treatment until death of any cause, patients who are still alive at their last follow-up will be censored at that time.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development
Locations (5):
- United States (5):
  - Desert Comprehensive Cancer Center, Palm Springs, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of North Carolina, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=330